CLINICAL TRIAL: NCT04454021
Title: Change in Muscle Volume in Patients With Unilateral Femoro-acetabular Impingement Syndrome After Hip Arthroscopy
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: wjqsportsmed163
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Femoro-acetabular Impingement (FAI)
Keywords: femoro-acetabular impingement; hip muscle volume; cross-sectional area; arthroscopy; MRI images
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hip arthroscopy — hip arthroscopy was performed when symptoms were not alleviated by nonsurgical treatment

SUMMARY:
The purpose of this study was to investigate the change in muscle volume around the hip in patients with unilateral femoro-acetabular impingement (FAI) after arthroscopy.

DETAILED DESCRIPTION:
We performed a retrospective review of magnetic resonance imaging (MRI) data of FAI patients who underwent hip arthroscopy between January 1, 2016, and July 1, 2018. "Image J" with an embedded region-of-interest (ROI) tool was used to calculate the cross-sectional area (CSA) of muscles on MRI. Wilcoxon signed-rank test was used to determine the differences between preoperative and postperative hip muscle CSA. The correlations of change in muscle CSA with age, gender, BMI, pain level, preoperative symptom duration, and multiple validated patient-reported outcomes were also analyzed with a spearman rank correlation test.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-50 years; (2) symptoms, physical examination, imaging evidence in accordance with FAI; (3) symptoms that were not alleviated by nonsurgical treatment; (4) the operation is performed by the same senior operator.

Exclusion Criteria:

* (1) bilateral symptoms; (2) revision surgery; (3) advanced osteoarthritis; (4) acetabular dysplasia; (5) history of hip and knee joint disease and operation; (6) osteonecrosis of hip; (7) sacroiliac joint disease

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: patients who underwent primary hip arthroscopy for the treatment of symptomatic FAI
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in muscle volume after hip arthroscopy | at least two years after hip arthroscopy
  hip muscle cross-sectional area of patients with unilateral FAI

CONTACTS AND LOCATIONS:
Locations (1):
- Jianquan Wang, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No